CLINICAL TRIAL: NCT05017844
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel Phase 2b/3 Study to Evaluate the Efficacy and Safety of KSR-001 in Patients With Dry Eye Syndrome
Brief Title: [KSR-001-P02] Phase 2b/3 Study, Evaluate the Efficacy and Safety of KSR-001 in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kukje Pharma (Other)
Collaborators: Samil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSR-001-P02
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KSR-001-04 (Placebo Comparator): KSR-001-04 eyedrops recieved one drop to both eyes four times a day for 12 weeks.
  Interventions: Drug: KSR-001-04
- KSR-001-02 (Experimental): KSR-001-02 eyedrops recieved one drop to both eyes four times a day for 12 weeks.
  Interventions: Drug: KSR-001-02
- KSR-001-03 (Experimental): KSR-001-03 eyedrops recieved one drop to both eyes four times a day for 12 weeks.
  Interventions: Drug: KSR-001-03

INTERVENTIONS:
Drug: KSR-001-04 — One drop to both eyes four times a day for 12 weeks
  Arms: KSR-001-04
Drug: KSR-001-02 — One drop to both eyes four times a day for 12 weeks
  Arms: KSR-001-02
Drug: KSR-001-03 — One drop to both eyes four times a day for 12 weeks
  Arms: KSR-001-03

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KSR-001 in patients with Dry Eye Syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female who over 19 years old
2. Those who have had symptoms of dry eye for at least 6 months (foreign body sensation, dryness, glare, pain pain, blurred vision, etc.) and Those whose symptoms do not improve with conservative treatment such as artificial tears
3. Those who meet below criteria at least one of two eyes

   * Those who have over than score 4 in corneal staining test
   * Tear secretion test without anesthesia(Schirmer test) result would be under 10mm/5min (If the test result is 0mm/5min, it should be over than 3mm/5min on the nasal stimulation schirmer test in the same eye)
4. both eyes, the corrected visual acuity is 0.2 or more
5. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. During this clinical trial period, When Rebamipide treatment is expected due to gastrointestinal disorder or gastritis
2. Within 90 days of the screening visit, if systemic steroid steroids or systemic immunosuppressants were used
3. Within 90 days of the screening visit, If there is a history of other ophthalmic surgeries including the use of punctum plugs or puncture closure surgery
4. If it is a clinically significant ophthalmic disease that is not caused by dry eye syndrome and may affect the interpretation of the results of this clinical trial
5. Within 90 days of the screening visit, Those who have undergone vision correction surgery such as LASIK or LASIK
6. Those with intraocular pressure (IOP) exceeding 21 mmHg or with glaucoma undergoing drug treatment
7. Those with hypersensitivity to the ingredient of this clinical trial drug
8. Patients planning to wear contact lenses during the clinical trial period
9. In the case of one of the following

   * Creatinine level more than twice the upper limit of normal range
   * AST or ALT levels greater than twice the upper limit of normal range
10. History of malignancy (except for cases where there has been no recurrence for more than 5 years after surgery)
11. Within 1 year before screening, Those who have been diagnosed with alcohol or drug abuse and are receiving treatment
12. In the case of women of childbearing potential, those who do not consent to contraception by a medically accepted method of contraception during the clinical trial period (IUD, Intrauterine device or IUS, Intrauterine system), tubal ligation, double blocking method (male condom, female condoms, cervical caps, contraceptive diaphragms, and Combination of blocking methods such as contraceptive sponges)
13. Pregnant or lactating women
14. within 30 days before participating in the clinical trial, Those who have applied other clinical trial drugs or medical devices
15. Patients judged by other investigators as unsuitable to participate in this clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Change in Fluorescein Corneal Staining (FCS) Score From Baseline to Last Observation Carried Forward (LOCF) | Baseline, 12 weeks
  FCS indicates the damage to the corneal epithelium. The degree of staining of the cornea after blue fluorescein staining under the slit lamp illumination of a cobalt blue light source was evaluated according to the National Eye Institute/Industry grading system.
  Per the National Eye Institute/Industry Workshop report, the cornea was divided into 5 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated(0-15)(0 is better).

SECONDARY OUTCOMES:
Fluorescein Corneal Staining (FCS) | Baseline, 4 weeks, 8 weeks
  The degree of staining of the cornea after blue fluorescein staining under the slit lamp illumination of a cobalt blue light source was evaluated according to the National Eye Institute/Industry grading system.
Lissamine Green Conjunctival Staining (LGCS) | Baseline, 4 weeks, 8 weeks, 12 weeks
  After lysamine green staining under slit lamps, the conjunctival staining was evaluated according to the National Eye Institute/Industry grading system.
Unanesthetized Schirmer's test | Baseline, 4 weeks, 8 weeks, 12 weeks
  After the eyes were wiped and the Schirmer test paper was inserted into the right eye at 1/3 of the lower eyelid without eye anesthesia and inserted into the left eye. After 5 minutes with the eyes closed, the Schirmer test paper was removed from the right side in the order of insertion and the left side removed. The wet length was measured in millimeters and the length of the midpoint was measured when the wet border was oblique.
Tear Film Break-up Time (TBUT) | Baseline, 4 weeks, 8 weeks, 12 weeks
  After blinking blue fluorescein staining of the cobalt blue light source, it was observed from the blinking point that there was a black spot, a streak pattern or a fluorine defect in the fluorescein-tear layer Was measured in seconds. The measurement results were repeated three times and average values were used.
Ocular Surface Disease Index (OSDI) | Baseline, 4 weeks, 8 weeks, 12 weeks
  The ocular surface disease index was assessed for ocular surface disease, including visual function (five items), eye symptoms (four items), and environmental factors (three items) , 0 point for none of the time, 1 point for some of the time, 2 points for half of the time, 3 points for most of the time, and 4 points for all of the time.

CONTACTS AND LOCATIONS:
Locations (1):
- Kukje Pharma, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No